CLINICAL TRIAL: NCT05971381
Title: The TONE Study: A Prospective Post-Market Clinical Study Investigating Repigmentation of Stable Vitiligo Lesions Using Spray-On Skin™ Cells
Brief Title: Repigmentation of Stable Vitiligo Lesions Using Spray-On Skin™ Cells
Acronym: TONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avita Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP010
Record Dates: First submitted 2023-07-24; First posted 2023-08-02 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Vitiligo
Keywords: focal vitiligo; segmental vitiligo; nonsegmental vitiligo; generalized vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Study Treatment (Other): Skin cell suspension prepared using the RECELL System will be applied to a prepared treatment area, followed by at-home NB-UVB phototherapy.
  Interventions: Device: RECELL® Autologous Cell Harvesting Device

INTERVENTIONS:
Device: RECELL® Autologous Cell Harvesting Device — The RECELL Device is for use at the patient's point-of-care for the safe and rapid preparation of Spray-On SkinTM Cells from a small sample of a patient's own skin.
  Other Names: Spray-On SkinTM Cells

SUMMARY:
To evaluate repigmentation and quality of life after treatment of stable vitiligo lesions using the RECELL Device.

DETAILED DESCRIPTION:
Prospective, multicenter single-arm pre-/post interventional study to evaluate the clinical performance of RECELL for repigmentation of stable depigmented lesions.Skin cell suspension prepared using the RECELL System will be applied to a prepared treatment area, followed by at-home NB-UVB phototherapy.

Repigmentation of treatment areas will be determined via centralized image interpretation by an expert dermatological panel (i.e., Central Review Committee, CRC).

ELIGIBILITY:
Inclusion Criteria:

1. Focal, segmental, or generalized (i.e., nonsegmental) stable vitiligo, defined as no new depigmented areas nor any depigmented areas that have expanded in size within the preceding 12 months.
2. The patient is a candidate for surgical intervention of a depigmented area, defined as a patient who has not satisfactorily responded to either:

   1. topical therapy or
   2. a minimum of 3 months of phototherapy.
3. The patient has a depigmented area available for treatment that is:

   1. ≥90% depigmented,
   2. without any other dermatologic conditions (other than vitiligo), and
   3. excludes the lips, eyelids, plantar surface of feet, palmar surface of hands.
4. The patient is 18 years of age or older.
5. The patient agrees to remain on any current use of immunosuppressive therapy for the duration of his/her participation in the study (52 weeks).
6. The patient is willing and able to comply with post-treatment at-home phototherapy and all follow-up study visits.
7. The patient agrees to abstain from any other treatment of the study area for the duration of his/her participation in the study (52 weeks).
8. The patient agrees to abstain from enrollment in any other interventional clinical trial for the duration of his/her participation in the study (52 weeks).
9. In the opinion of the investigator, the patient must be able to:

   1. Understand the full nature and purpose of the study, including possible risks and benefits,
   2. Understand instructions and be able to comprehend and complete study questionnaires, and
   3. Provide voluntary written informed consent. -

Exclusion Criteria:

1. The patient is unable to undergo treatment area preparation.
2. Patients who received RECELL treatment for vitiligo in Protocol No. CTP008 or CTP009.
3. Patients with:

   1. depigmented lips and fingertips (lip-tip vitiligo), or
   2. depigmented areas over >30% of their body surface area.
4. Patients with recent history (within previous 12 months) of:

   1. Koebnerization,
   2. confetti-like, or
   3. trichrome lesions.
5. Patients with a history of keloid formation.
6. The patient has other concurrent conditions that in the opinion of the investigator may compromise patient safety or study objectives.
7. Current use of medications (e.g., anticoagulants such as heparin or warfarin) that in the investigator's opinion may compromise patient safety or trial objectives.
8. The patient has a known hypersensitivity to trypsin, compound sodium lactate for irrigation solution (Hartmann's solution), povidone-iodine, chlorhexidine, and/or lidocaine-containing anesthetics -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Repigmentation 0%,1-25%, 26-50%, 51-79%, 80-99%, and 100%) | 24 weeks post-treatment
  Central Review Committee categorization of index area repigmentation

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Affiliated Dermatology, Scottsdale, Arizona
  - University of California, Irvine, Irvine, California
  - West Dermatology Research Center, San Diego, California
  - Sutter Health, Sunnyvale, California
  - California Dermatology Institute, Thousand Oaks, California
  - Clarity Dermatology, Castle Rock, Colorado
  - Siperstein Dermatology Group, Boynton Beach, Florida
  - Skin Care Research, LLC, Hollywood, Florida
  - Dermatologic Surgery Center of Washington, Chevy Chase, Maryland
  - Maryland Laser, Skin & Vein Institute, Hunt Valley, Maryland
  - University Of Massachusetts, Worcester, Massachusetts
  - Hamzavi Dermatology, Canton, Michigan
  - Henry Ford Health, Detroit, Michigan
  - Grekin Skin Institute, Warren, Michigan
  - The Dermatology Specialist, New York, New York
  - Mount Sinai, New York, New York
  - Dermatology, Laser and Vein Specialists of the Carolinas, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No